CLINICAL TRIAL: NCT04244630
Title: Mitochondrial Capacity Boost in ALS (MICABO-ALS) Trial
Acronym: MICABO-ALS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-094
Record Dates: First submitted 2020-01-22; First posted 2020-01-28 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Antioxidants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Antioxidants (Other): Eligible patients will receive over-the-counter anti-oxidants, namely vitamin E, NAc cysteine, L-cystine, Nicotinamide and Taurursodiol at defined doses.
  Interventions: Combination Product: Antioxidants

INTERVENTIONS:
Combination Product: Antioxidants — Over-the-counter anti-oxidants, namely vitamin E, NAc cysteine, L-cystine, Nicotinamide and Taurursodiol at defined doses

SUMMARY:
The purpose of this research is to investigate the validity of a previous clinical trial named EH301, which showed beneficial effects of anti-oxidant therapies in patients with amyotrophic lateral sclerosis (ALS). If validated by this study, providing over-the-counter anti-oxidants would be a simple, low risk, low-cost approach to significantly slow or stop the progression of ALS, for which currently no effective treatment exists. It is currently thought that oxidative stress is a major cause of ALS. The study investigators are therefore planning to expand the original scope of the previous trial by including anti-oxidants at high doses that were not previously used. All of these compounds are considered safe.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disorder that affects muscle function throughout the body. Weakness and muscle shrinkage begin either in the face, arm, or leg. A clinical ALS hallmark is rapidly progressive weight loss. Also, respiration is usually affected late in the disease, and death typically occurs as a consequence of respiratory failure. The median survival after disease onset is approximately 3-4 years.

While there are now two FDA-approved agents for patients with ALS, there are no interventions that have had a meaningful impact on the natural course of this disease. Riluzole prolongs survival by up to 12 weeks. Edaravone improves some aspects of neurological function in a small subset of patients, but that was ineffective in clinical studies that included ALS patients at all stages of disease.

Past failures to identify effective therapies reflect the complexity of ALS pathogenesis, in that no single therapeutic target has been identified. Thus, single agent or dual combination therapies are unlikely to succeed. Given the truly rapid and devastating nature of ALS and that there are no effective treatments for ALS, one can argue that it is critical to devise a different approach. Until the exact mechanisms that lead to ALS are identified, it is necessary to employ polytherapy which includes new agents that show promise.

This study will lay further groundwork on methodology for performing more definite trials in ALS. The study of secondary biomarkers in ALS is significant because there are currently no molecular or biochemical biomarkers for assessing therapeutic efficacy of drug treatments in ALS clinical trials. By doing this study, the study investigators hope to learn that high-dose anti-oxidants would be a simple, low risk, low-cost approach to significantly slow or stop the progression of ALS, for which currently no effective treatment exists. Participation in this research will last about 13 months

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis by a study investigator of laboratory-supported probable, probable, or definite ALS, according to a modified El Escorial criterion (Appendix 2).
2. 21 to 80 years of age inclusive.
3. If patients are taking riluzole for ALS, they must be on a stable dose for at least thirty days prior to the baseline visit.
4. Willing and able to give signed informed consent that has been approved by the Institutional Review Board (IRB).

Exclusion Criteria:

1. Diagnosis of other neurodegenerative diseases (Parkinson disease, Alzheimer disease, etc.).
2. Clinically significant history of unstable medical illness (unstable angina, advanced cancer, etc.) over the last 30 days.
3. Infection with the human immunodeficiency virus (HIV)
4. Limited mental capacity such that the patient cannot provide written informed consent or comply with evaluation procedures.
5. History of recent alcohol or drug abuse or noncompliance with treatment or other experimental protocols. 6 Receipt of any investigational drug within the past 30 days.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of serum NfL | 12 months
  The change in log serum NfL level from baseline to 12 months will be assessed using a linear mixed model and the differences in NfL level at 12 months from baseline assessed using a paired t-test.

SECONDARY OUTCOMES:
Measurement of functional decline in ALS | 12 months
  Functional decline in ALS patients will be measured using the ALS Functional Rating Scale - Revised (ALSFRS-R), change will be measured from baseline to 12 months.
  The ALSFRS-R is a quickly administered (five minutes) ordinal rating scale that assesses patients' capability and independence in 12 functional activities.
Frequency of serious adverse events and adverse events. | 12 months
  The frequency of serious adverse events and adverse events will be summarized using frequency and percentages.
Survival analysis | 12 months
  This is a robust measure of effect in this rapidly progressing terminal disease. Survival has been a standard outcome measure in past clinical trials.

OTHER OUTCOMES:
Change in serum CK level from baseline to 12 months | 12 months
  CK levels will be measured in a clinical laboratory by colorimetric measurements. Analysis of serum CK levels will be conducted similar to serum NfL.

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Stuve, M.D., Ph.D., Principal Investigator — Dallas VA Medical Center
Locations (1):
- VA North Texas Health Care System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rowland LP, Shneider NA. Amyotrophic lateral sclerosis. N Engl J Med. 2001 May 31;344(22):1688-700. doi: 10.1056/NEJM200105313442207. No abstract available. PMID 11386269
- [Background] Akao Y, Maruyama W, Shimizu S, Yi H, Nakagawa Y, Shamoto-Nagai M, Youdim MB, Tsujimoto Y, Naoi M. Mitochondrial permeability transition mediates apoptosis induced by N-methyl(R)salsolinol, an endogenous neurotoxin, and is inhibited by Bcl-2 and rasagiline, N-propargyl-1(R)-aminoindan. J Neurochem. 2002 Aug;82(4):913-23. doi: 10.1046/j.1471-4159.2002.01047.x. PMID 12358797
- [Background] O'Toole O, Traynor BJ, Brennan P, Sheehan C, Frost E, Corr B, Hardiman O. Epidemiology and clinical features of amyotrophic lateral sclerosis in Ireland between 1995 and 2004. J Neurol Neurosurg Psychiatry. 2008 Jan;79(1):30-2. doi: 10.1136/jnnp.2007.117788. Epub 2007 Jul 18. PMID 17634215
- [Background] Logroscino G, Traynor BJ, Hardiman O, Chio A, Mitchell D, Swingler RJ, Millul A, Benn E, Beghi E; EURALS. Incidence of amyotrophic lateral sclerosis in Europe. J Neurol Neurosurg Psychiatry. 2010 Apr;81(4):385-90. doi: 10.1136/jnnp.2009.183525. Epub 2009 Aug 25. PMID 19710046
- [Background] Huisman MH, de Jong SW, van Doormaal PT, Weinreich SS, Schelhaas HJ, van der Kooi AJ, de Visser M, Veldink JH, van den Berg LH. Population based epidemiology of amyotrophic lateral sclerosis using capture-recapture methodology. J Neurol Neurosurg Psychiatry. 2011 Oct;82(10):1165-70. doi: 10.1136/jnnp.2011.244939. Epub 2011 May 27. PMID 21622937
- [Background] Wittie M, Nelson LM, Usher S, Ward K, Benatar M. Utility of capture-recapture methodology to assess completeness of amyotrophic lateral sclerosis case ascertainment. Neuroepidemiology. 2013;40(2):133-41. doi: 10.1159/000342156. Epub 2012 Oct 24. PMID 23095852
- [Background] van Es MA, Hardiman O, Chio A, Al-Chalabi A, Pasterkamp RJ, Veldink JH, van den Berg LH. Amyotrophic lateral sclerosis. Lancet. 2017 Nov 4;390(10107):2084-2098. doi: 10.1016/S0140-6736(17)31287-4. Epub 2017 May 25. PMID 28552366
- [Background] Brooks BR. El Escorial World Federation of Neurology criteria for the diagnosis of amyotrophic lateral sclerosis. Subcommittee on Motor Neuron Diseases/Amyotrophic Lateral Sclerosis of the World Federation of Neurology Research Group on Neuromuscular Diseases and the El Escorial "Clinical limits of amyotrophic lateral sclerosis" workshop contributors. J Neurol Sci. 1994 Jul;124 Suppl:96-107. doi: 10.1016/0022-510x(94)90191-0. No abstract available. PMID 7807156
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847
- [Background] Gubbay SS, Kahana E, Zilber N, Cooper G, Pintov S, Leibowitz Y. Amyotrophic lateral sclerosis. A study of its presentation and prognosis. J Neurol. 1985;232(5):295-300. doi: 10.1007/BF00313868. PMID 4056836
- [Background] Eisen A, Schulzer M, MacNeil M, Pant B, Mak E. Duration of amyotrophic lateral sclerosis is age dependent. Muscle Nerve. 1993 Jan;16(1):27-32. doi: 10.1002/mus.880160107. PMID 8423829
- [Background] Taylor JP, Brown RH Jr, Cleveland DW. Decoding ALS: from genes to mechanism. Nature. 2016 Nov 10;539(7628):197-206. doi: 10.1038/nature20413. PMID 27830784
- [Background] Hokkanen SRK, Hunter S, Polvikoski TM, Keage HAD, Minett T, Matthews FE, Brayne C; MRC CFAS and CC75C Study Group. Hippocampal sclerosis, hippocampal neuron loss patterns and TDP-43 in the aged population. Brain Pathol. 2018 Jul;28(4):548-559. doi: 10.1111/bpa.12556. Epub 2017 Sep 25. PMID 28833898
- [Background] Keage HA, Hunter S, Matthews FE, Ince PG, Hodges J, Hokkanen SR, Highley JR, Dening T, Brayne C. TDP-43 pathology in the population: prevalence and associations with dementia and age. J Alzheimers Dis. 2014;42(2):641-50. doi: 10.3233/JAD-132351. PMID 25170584
- [Background] Neumann M, Sampathu DM, Kwong LK, Truax AC, Micsenyi MC, Chou TT, Bruce J, Schuck T, Grossman M, Clark CM, McCluskey LF, Miller BL, Masliah E, Mackenzie IR, Feldman H, Feiden W, Kretzschmar HA, Trojanowski JQ, Lee VM. Ubiquitinated TDP-43 in frontotemporal lobar degeneration and amyotrophic lateral sclerosis. Science. 2006 Oct 6;314(5796):130-3. doi: 10.1126/science.1134108. PMID 17023659
- [Background] Doble A. The pharmacology and mechanism of action of riluzole. Neurology. 1996 Dec;47(6 Suppl 4):S233-41. doi: 10.1212/wnl.47.6_suppl_4.233s. PMID 8959995
- [Background] Cruz MP. Edaravone (Radicava): A Novel Neuroprotective Agent for the Treatment of Amyotrophic Lateral Sclerosis. P T. 2018 Jan;43(1):25-28. PMID 29290672
- [Background] de la Rubia JE, Drehmer E, Platero JL, Benlloch M, Caplliure-Llopis J, Villaron-Casales C, de Bernardo N, AlarcOn J, Fuente C, Carrera S, Sancho D, GarcIa-Pardo P, Pascual R, JuArez M, Cuerda-Ballester M, Forner A, Sancho-Castillo S, Barrios C, Obrador E, Marchio P, Salvador R, Holmes HE, Dellinger RW, Guarente L, Estrela JM. Efficacy and tolerability of EH301 for amyotrophic lateral sclerosis: a randomized, double-blind, placebo-controlled human pilot study. Amyotroph Lateral Scler Frontotemporal Degener. 2019 Feb;20(1-2):115-122. doi: 10.1080/21678421.2018.1536152. Epub 2019 Jan 22. PMID 30668199
- [Background] Yin TC, Britt JK, De Jesus-Cortes H, Lu Y, Genova RM, Khan MZ, Voorhees JR, Shao J, Katzman AC, Huntington PJ, Wassink C, McDaniel L, Newell EA, Dutca LM, Naidoo J, Cui H, Bassuk AG, Harper MM, McKnight SL, Ready JM, Pieper AA. P7C3 neuroprotective chemicals block axonal degeneration and preserve function after traumatic brain injury. Cell Rep. 2014 Sep 25;8(6):1731-1740. doi: 10.1016/j.celrep.2014.08.030. Epub 2014 Sep 15. PMID 25220467
- [Background] Pieper M, Scheffold C, Duwe S, Rossig C, Bisping G, Stelljes M, Tedder TF, Jurgens H, Berdel WE, Kienast J. Immunotherapy of B-cell malignancies with genetically engineered human CD8+ natural killer T cells. Leukemia. 2006 Apr;20(4):729-32. doi: 10.1038/sj.leu.2404114. No abstract available. PMID 16437143
- [Background] Wang G, Han T, Nijhawan D, Theodoropoulos P, Naidoo J, Yadavalli S, Mirzaei H, Pieper AA, Ready JM, McKnight SL. P7C3 neuroprotective chemicals function by activating the rate-limiting enzyme in NAD salvage. Cell. 2014 Sep 11;158(6):1324-1334. doi: 10.1016/j.cell.2014.07.040. PMID 25215490
- [Background] Evers BM, Rodriguez-Navas C, Tesla RJ, Prange-Kiel J, Wasser CR, Yoo KS, McDonald J, Cenik B, Ravenscroft TA, Plattner F, Rademakers R, Yu G, White CL 3rd, Herz J. Lipidomic and Transcriptomic Basis of Lysosomal Dysfunction in Progranulin Deficiency. Cell Rep. 2017 Sep 12;20(11):2565-2574. doi: 10.1016/j.celrep.2017.08.056. PMID 28903038
- [Background] Radford RA, Morsch M, Rayner SL, Cole NJ, Pountney DL, Chung RS. The established and emerging roles of astrocytes and microglia in amyotrophic lateral sclerosis and frontotemporal dementia. Front Cell Neurosci. 2015 Oct 27;9:414. doi: 10.3389/fncel.2015.00414. eCollection 2015. PMID 26578880
- [Background] Desai VG, Herman EH, Moland CL, Branham WS, Lewis SM, Davis KJ, George NI, Lee T, Kerr S, Fuscoe JC. Development of doxorubicin-induced chronic cardiotoxicity in the B6C3F1 mouse model. Toxicol Appl Pharmacol. 2013 Jan 1;266(1):109-21. doi: 10.1016/j.taap.2012.10.025. Epub 2012 Nov 7. PMID 23142469
- [Background] Gaiottino J, Norgren N, Dobson R, Topping J, Nissim A, Malaspina A, Bestwick JP, Monsch AU, Regeniter A, Lindberg RL, Kappos L, Leppert D, Petzold A, Giovannoni G, Kuhle J. Increased neurofilament light chain blood levels in neurodegenerative neurological diseases. PLoS One. 2013 Sep 20;8(9):e75091. doi: 10.1371/journal.pone.0075091. eCollection 2013. PMID 24073237
- [Background] Lu CH, Macdonald-Wallis C, Gray E, Pearce N, Petzold A, Norgren N, Giovannoni G, Fratta P, Sidle K, Fish M, Orrell R, Howard R, Talbot K, Greensmith L, Kuhle J, Turner MR, Malaspina A. Neurofilament light chain: A prognostic biomarker in amyotrophic lateral sclerosis. Neurology. 2015 Jun 2;84(22):2247-57. doi: 10.1212/WNL.0000000000001642. Epub 2015 May 1. PMID 25934855
- [Background] Benatar M, Wuu J, Andersen PM, Lombardi V, Malaspina A. Neurofilament light: A candidate biomarker of presymptomatic amyotrophic lateral sclerosis and phenoconversion. Ann Neurol. 2018 Jul;84(1):130-139. doi: 10.1002/ana.25276. Epub 2018 Aug 16. PMID 30014505
- [Background] Verde F, Steinacker P, Weishaupt JH, Kassubek J, Oeckl P, Halbgebauer S, Tumani H, von Arnim CAF, Dorst J, Feneberg E, Mayer B, Muller HP, Gorges M, Rosenbohm A, Volk AE, Silani V, Ludolph AC, Otto M. Neurofilament light chain in serum for the diagnosis of amyotrophic lateral sclerosis. J Neurol Neurosurg Psychiatry. 2019 Feb;90(2):157-164. doi: 10.1136/jnnp-2018-318704. Epub 2018 Oct 11. PMID 30309882
- [Background] Thouvenot E, Demattei C, Lehmann S, Maceski-Maleska A, Hirtz C, Juntas-Morales R, Pageot N, Esselin F, Alphandery S, Vincent T, Camu W. Serum neurofilament light chain at time of diagnosis is an independent prognostic factor of survival in amyotrophic lateral sclerosis. Eur J Neurol. 2020 Feb;27(2):251-257. doi: 10.1111/ene.14063. Epub 2019 Sep 18. PMID 31437330
- [Background] Feneberg E, Oeckl P, Steinacker P, Verde F, Barro C, Van Damme P, Gray E, Grosskreutz J, Jardel C, Kuhle J, Koerner S, Lamari F, Amador MDM, Mayer B, Morelli C, Muckova P, Petri S, Poesen K, Raaphorst J, Salachas F, Silani V, Stubendorff B, Turner MR, Verbeek MM, Weishaupt JH, Weydt P, Ludolph AC, Otto M. Multicenter evaluation of neurofilaments in early symptom onset amyotrophic lateral sclerosis. Neurology. 2018 Jan 2;90(1):e22-e30. doi: 10.1212/WNL.0000000000004761. Epub 2017 Dec 6. PMID 29212830
- [Background] Kaufmann P, Levy G, Montes J, Buchsbaum R, Barsdorf AI, Battista V, Arbing R, Gordon PH, Mitsumoto H, Levin B, Thompson JL; QALS study group. Excellent inter-rater, intra-rater, and telephone-administered reliability of the ALSFRS-R in a multicenter clinical trial. Amyotroph Lateral Scler. 2007 Feb;8(1):42-6. doi: 10.1080/17482960600888156. PMID 17364435
- [Background] Cudkowicz M, Bozik ME, Ingersoll EW, Miller R, Mitsumoto H, Shefner J, Moore DH, Schoenfeld D, Mather JL, Archibald D, Sullivan M, Amburgey C, Moritz J, Gribkoff VK. The effects of dexpramipexole (KNS-760704) in individuals with amyotrophic lateral sclerosis. Nat Med. 2011 Nov 20;17(12):1652-6. doi: 10.1038/nm.2579. PMID 22101764